CLINICAL TRIAL: NCT02737332
Title: A Randomized, Open-Label, Active-Controlled, Multi-Center Study to Evaluate Serum Testosterone Levels in Patients With Metastatic Castration-Resistant Prostate Cancer: The STAAR STUDY
Brief Title: A Study to Evaluate Serum Testosterone Levels in Patients With Metastatic Castration-Resistant Prostate Cancer
Acronym: STAAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHL-AA-201
Record Dates: First submitted 2016-03-25; First posted 2016-04-13 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zytiga® (Abiraterone Acetate) (Active Comparator): 1,000 MG (4 x 250 mg qd)
  Interventions: Drug: Zytiga® (Abiraterone Acetate)
- SoluMatrix™ (Abiraterone Acetate) (Experimental): 500 mg (4 x 125 mg qd)
  Interventions: Drug: SoluMatrix™ (Abiraterone Acetate)

INTERVENTIONS:
Drug: Zytiga® (Abiraterone Acetate) — Zytiga® 1,000 mg (4 x 250 mg qd) tablets plus one 5 mg prednisone tablet to be taken bid, spaced approximately 12 hours apart
  Other Names: Zytiga®
  Arms: Zytiga® (Abiraterone Acetate)
Drug: SoluMatrix™ (Abiraterone Acetate) — SoluMatrix™ 500 mg (4 x 125 mg qd) tablets plus one 4 mg methylprednisolone tablet bid, spaced approximately 12 hours apart
  Other Names: SoluMatrix™
  Arms: SoluMatrix™ (Abiraterone Acetate)

SUMMARY:
The purpose of this study is to evaluate the serum testosterone levels in patients with Metastatic Castration-Resistant Prostate Cancer on SoluMatrix™ Abiraterone Acetate as Compared to Abiraterone Acetate

DETAILED DESCRIPTION:
This was a 12-week, open-label study of abiraterone acetate in at least 50 patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed
2. Male subjects at least 18 years of age or older at time of consent
3. Pathologically confirmed adenocarcinoma of the prostate
4. Ongoing therapy with a GnRH agonist or antagonist AND serum testosterone level <50 ng/dL at screening
5. Metastatic disease documented by computed tomography (CT)/ magnetic resonance imaging (MRI) or bone scan. Imaging obtained within 42 days prior to the start of study medication will be accepted.
6. Meeting disease progression according to the recommendations of the prostate cancer working group 2 by one of the following criteria:

   * Two rises of PSA (taken a minimum of 1 week apart) from a baseline measurement of at least 2 ng/mL,
   * Imaging progression (CT/MRI) by RECIST criteria
   * Nuclear scan progression by new lesion.
7. Discontinuation of flutamide or nilutamide, and other anti-androgens at least 4 weeks prior to the start of study medication; discontinuation of bicalutamide at least 6 weeks prior to start of study medication.
8. Discontinuation of Radiotherapy > 4 weeks prior to start of study medication.
9. ECOG performance status of 0-1 at screening
10. Screening blood counts of the following:

    * Absolute neutrophil count > 1500/µL
    * Platelets > 100,000/µL
    * Hemoglobin > 9 g/dL
11. Screening chemistry values of the following:

    * ALT and AST < 2.5 x ULN
    * Total bilirubin < 1.5 x ULN
    * Creatinine< 1.5 x ULN
    * Albumin > 3.0 g/dL
12. Potassium > 3.5 mmol/L
13. Life expectancy of at least 6 months at screening
14. Subject is willing and able to comply with all protocol requirements assessments
15. Agrees to protocol-defined use of effective contraception.

Exclusion Criteria:

1. History of impaired pituitary or adrenal gland function
2. Prior therapy with abiraterone acetate, orteronel, ketoconazole or any other CYP17 inhibitor
3. Prior therapy with enzalutamide
4. Prior use of experimental androgen receptor antagonist
5. Previous exposure to Ra-223:Xofigo
6. Previous chemotherapy
7. Initiation of bisphosphonate or denosumab therapy within 30 days prior to the start of study medication. Patients who are on a stable dose of these medications for at least 30 days at the time of starting study drug are eligible.
8. Therapy with estrogen within 30 days prior to the start of study medication
9. Use of systemic glucocorticoids equivalent to > 10 mg of prednisone daily; patients who have discontinued or have reduced dose to < 10 mg prednisone within 14 days prior to the start of study medication will be eligible
10. Prior use of any herbal products that may decrease PSA levels (eg., saw palmetto) within 30 days of start of study medication
11. Known metastases to the brain or CNS involvement
12. History of other malignancy within the previous 2 years
13. Major surgery within 30 days prior to the start of study medication
14. Blood transfusion within 30 days of screening
15. Serious, persistent infection within 14 days of the start of study medication
16. Persistent pain that requires the use of a narcotic analgesic
17. Known gastrointestinal disease or condition that may impair absorption
18. Treatment with any investigational drug within 4 weeks prior to Day -1 of the study.
19. Known history of human immunodeficiency virus (HIV) or seropositive test for hepatitis C virus or hepatitis B virus
20. Have poorly controlled diabetes.
21. Uncontrolled hypertension
22. History of New York Heart Association (NYHA) class III or IV heart failure
23. Serious concurrent illness, including psychiatric illness, that would interfere with study participation
24. Inability to swallow tablets whole
25. Known hypersensitivity to any excipients in study medications
26. Moderate to severe hepatic impairment (Child-Pugh Classes B and C)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nemeth, PhD, Study Director
Locations (17):
- United States (17):
  - Alliance Research, Laguna Hills, California
  - Tower Urology, Los Angeles, California
  - San Bernardino Urological, San Bernardino, California
  - Skyline Urology, Torrance, California
  - Innovative Clinical Research Institute, Whittier, California
  - Urology Associates, P.C., Englewood, Colorado
  - Manatee Medical Research, Bradenton, Florida
  - North Idaho Urology, Coeur d'Alene, Idaho
  - The Iowa Clinic, West Des Moines, Iowa
  - Wichita Urology Group, Wichita, Kansas
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Lincoln Urology, PC, Lincoln, Nebraska
  - Urology Cancer Center, Omaha, Nebraska
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Associated Urologist of North Carolina, Raleigh, North Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zytiga® (Abiraterone Acetate): Zytiga® 1,000 mg (4 x 250 mg qd) tablets
- SoluMatrix™ (Abiraterone Acetate): SoluMatrix™ 500 mg (4 x 125 mg qd) tablets
Period: Overall Study
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Started | 29 | 24
Completed | 28 | 23
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate) | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (9.4) | 77 (8.9) | 75.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 24 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 27 | 20 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 24 | 53

OUTCOME MEASURES:

1. Primary Outcome: Testosterone Levels
Description: Blood Sample tested for Serum Testosterone Levels
Time Frame: Average of Day 9 and 10
Population: Analysis of serum T levels in the ITT population
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 29 | 24
ng/dL | 1.02 (0.03) | 1.05 (0.04)
Statistical Analysis 1: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Equivalence — The bioequivalence between the two products was concluded if the 90% CIs (based on log transformed data and anti-logged) for the ratio of the geometric means lie completely within the range 80%-125%; p = 0.4879, ANOVA — One-way ANOVA model with treatment as the independent variable, and the least-square means and standard error of Testosterone levels under each treatment and the between-treatment difference in LS means was reported; Geometric mean ratio of treatments = 1.019, 90% CI 2-sided [0.964 to 1.077] — Geometric mean ratio of experimental and reference product was determined by exponentiating least-squares means of log-transformed value

2. Secondary Outcome: PSA Levels
Description: All patients randomized to one of the two treatment groups, round about level of PSA.
  These were assessed only at the said Outcome Measure Time Frame. No additional time points to the said endpoint
Time Frame: Day 28, Day 56, and Day 84
Population: ITT population:The intention-to-treat (ITT) population is defined as all subjects who are randomized to one of the two treatment groups. The ITT population is the primary population for PD evaluation. The ITT population will be identified and finalized before the database is locked.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 29 | 24
ng/mL
  Day 28 | 37.5 (11.33) | 22.37 (12.02)
  Day 56 | 40.84 (12.58) | 25.29 (13.68)
  Day 84 | 33.88 (13.43) | 26.46 (15.41)
Statistical Analysis 1: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3642, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio = 0.994, 90% CI 2-sided [0.0451 to 2.192] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4069, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio = 0.810, 90% CI 2-sided [0.338 to 1.939] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Equivalence — One-way ANOVA model with treatment as the independent variable, and the least-square means and standard error of Testosterone levels under each treatment and the between-treatment difference in LS means was reported; p = 0.7186, ANOVA — The bioequivalence between the two products was concluded if the 90% CIs (based on log transformed data and anti-logged) for the ratio of the geometric means lie completely within the range 80%-125%; Geometric mean ratio = 1.039, 90% CI 2-sided [0.412 to 2.617] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percent of Subjects With PSA-50 Response
Description: Proportion of patients with complete suppression of PSA-50 were reported by treatment and compared for between-group differences.
  These were assessed only at the said Outcome Measure Time Frame. No additional time points to the said endpoint.
Time Frame: Day 28, Day 56, and Day 84
Population: as for outcome 2
Measure: Number; unit: percentage of Participants
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 27 | 24
percentage of Participants
  Day 28 | 70.4 | 66.7
  Day 56: number analyzed (Participants) | 26 | 22
  Day 56 | 65.4 | 63.6
  Day 84: number analyzed (Participants) | 25 | 19
  Day 84 | 72.0 | 68.4
Statistical Analysis 1: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Other; p = 1.0000, Fisher Exact

4. Secondary Outcome: Serum Testosterone Levels
Description: These were assessed only at the said Outcome Measure Time Frame. No additional time points to the said endpoint.
Time Frame: Day 28, Day 56, and Day 84
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 29 | 24
ng/dL
  Day 28 | 1.01 (0.01) | 1.01 (0.01)
  Day 56 | 1.01 (1.03) | 2.56 (1.07)
  Day 84 | 1 (0) | 1 (0)
Statistical Analysis 1: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9211, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio = 0.999, 90% CI 2-sided [0.980 to 1.018] — [estimate comment as in outcome 1, analysis 1]; ANOVA-model-based Least-Square Mean
Statistical Analysis 2: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3037, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.168, 90% CI 2-sided [0.900 to 1.515] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.000, 90% CI 2-sided [1.000 to 1.000] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Steady State Trough Concentration of Arbiraterone
Description: These were assessed only at the said Outcome Measure Time Frame. No additional time points to the said endpoint.
Time Frame: Day 09, Day 28, Day 56, and Day 84
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 28 | 23
ng/dL
  Day 09 | 20.938 (7.044) | 27.259 (7.772)
  Day 28: number analyzed (Participants) | 23 | 21
  Day 28 | 56.721 (23.104) | 18.662 (24.18)
  Day 56: number analyzed (Participants) | 23 | 18
  Day 56 | 29.978 (8.117) | 18.707 (9.175)
  Day 84: number analyzed (Participants) | 18 | 15
  Day 84 | 18.263 (3.087) | 13.819 (3.381)
Statistical Analysis 1: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Other; p = 0.5495, ANOVA
Statistical Analysis 2: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Other; p = 0.2616, ANOVA
Statistical Analysis 3: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Other; p = 0.3632, ANOVA
Statistical Analysis 4: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Other; p = 0.3393, ANOVA

6. Secondary Outcome: AUC (0-inf)
Description: Steady state systemic exposure parameters
Time Frame: 60 to 30 minutes prior to dosing and over 24 Hours post-dose
Measure: Least Squares Mean (Standard Error); unit: ng*hr/mL
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 8 | 4
ng*hr/mL | 1020.218 (154.549) | 326.458 (218.565)

7. Secondary Outcome: AUC (0-24 hr)
Description: Blood samples for pre-dose PK profiling were to be collected approximately 45 minutes before dosing, i.e., within 60 to 30 minutes prior to dosing. Post-dose blood samples were to be collected throughout the day at the times (15 mins, 30 mins, 1 hr, 1.5 hr, 2.0 hr 3 hr, 4 hr, 6 hr, 8 hr, 9 hr, 24 hr).
Time Frame: 60 to 30 minutes prior to dosing and over 24 Hours post-dose
Population: Overall, 14 subjects were analyzed in the PK population, amongst which, 8 were in the Zytiga group and 5 were in the SoluMatrix group.
Measure: Least Squares Mean (Standard Error); unit: ng*hr/mL
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 8 | 5
ng*hr/mL | 870.859 (221.709) | 626.066 (280.443)

8. Secondary Outcome: AUC (0-t)
Description: as for outcome 7
Time Frame: 60 to 30 minutes prior to dosing and over 24 Hours post-dose
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: ng*hr/mL
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 8 | 5
ng*hr/mL | 870.859 (221.709) | 626.066 (280.443)

9. Secondary Outcome: Cmax
Description: as for outcome 7
Time Frame: 60 to 30 minutes prior to dosing and over 24 Hours post-dose
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Groups:
- SoluMatrix™ (Abiraterone Acetate): 500 mg (4 x 125 mg qd)
  SoluMatrix™ (Abiraterone Acetate): SoluMatrix™ Abiraterone Acetate 500 mg Compared to Zytiga® 1,000 mg (4 x 250 mg qd)
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
Number analyzed (Participants) | 8 | 5
ng/mL | 268.261 (69.967) | 111.316 (88.503)
Statistical Analysis 1: Comparison: Zytiga® (Abiraterone Acetate) vs SoluMatrix™ (Abiraterone Acetate); Test type: Other; p = 0.1917, ANOVA

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of signing of the ICF until study completion (84 Days). The AEs collected in the source documents for screening failures did not need to be entered into eCRF, however once a potential patient was randomized, all AEs were to be entered into the eCRF.
Description: The investigator monitored and/or asked about or evaluated AEs using non-leading questions at each visit or evaluation.
Groups:
- Zytiga® (Abiraterone Acetate): 1,000 MG (4 x 250 mg qd)
  Zytiga® (Abiraterone Acetate): Zytiga® 1,000 mg (4 x 250 mg qd) Compared to SoluMatrix™ Abiraterone Acetate 500 mg
Arm/Group | Zytiga® (Abiraterone Acetate) | SoluMatrix™ (Abiraterone Acetate)
All-Cause Mortality (participants affected / at risk) | 2/29 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/29 | 5/24
Other Adverse Events (participants affected / at risk) | 22/29 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zytiga® (Abiraterone Acetate) (N=29) | SoluMatrix™ (Abiraterone Acetate) (N=24)
Corornary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Progression of prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Infections and infestations) | 0 (0) | 1 (1)
Worsening of left hydroureteronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zytiga® (Abiraterone Acetate) (N=29) | SoluMatrix™ (Abiraterone Acetate) (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Urinary tract infections (Infections and infestations) | 3 | 4
Blood creatiineincreased (Investigations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 4 | 0
Hypertension (Vascular disorders) | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Gastroesophgeal reflux disease (Gastrointestinal disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT02737332/Prot_SAP_000.pdf